CLINICAL TRIAL: NCT01208233
Title: A Phase 2 Multicenter, Randomized, Double Blind, Placebo Controlled Study Of The Safety And Efficacy Of Pf-03049423 In Subjects With Ischemic Stroke
Brief Title: Study Evaluating The Safety And Efficacy Of PF-03049423 In Subjects With Ischemic Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9541004; 2010-021414-32 (EudraCT Number)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Ischemic Stroke
Keywords: Phase 2 Ischemic stroke Safety and efficacy
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-(4-(2-hydroxyethyl)piperazin-1-yl)-7-(6-methoxypyridin-3-yl)-1-(2-propoxyethyl)pyrido(3,4-b)pyrazin-2(1H)-one

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 mg PF-03049423 (Experimental)
  Interventions: Drug: PF-03049423
- 3 mg of PF-03049423 (Experimental)
  Interventions: Drug: PF-03049423
- 6 mg of PF-03049423 (Experimental)
  Interventions: Drug: PF-03049423
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-03049423 — 1 mg of PF-03049423 daily for 90 days
  Arms: 1 mg PF-03049423
Drug: PF-03049423 — 3 mg of PF-03049423 daily for 90 days
  Arms: 3 mg of PF-03049423
Drug: PF-03049423 — 6 mg of PF-03049423 daily for 90 days
  Arms: 6 mg of PF-03049423
Other: Placebo — Placebo of PF-03049423 daily for 90 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of PF-03049423 following multiple dose administration to subjects with ischemic stroke. The study will also evaluate the efficacy of PF-03049423, relative to placebo, in subjects with ischemic stroke following 90 days of therapy. The study will also explore the relationship between PF-03049423 concentration and blood pressure.

DETAILED DESCRIPTION:
The interim analysis for the POC study A9541004 demonstrated futility, and the study was stopped on the 6th of November 2013. There were no signals of serious safety concern.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic stroke with an onset within 72 hours prior to start of study agent administration, male or female.
* Supratentorial ischemic stroke involving the cortex documented by neurological exam and confirmed by MRI.
* Stroke involving upper extremity.
* Subjects who received thrombolytic therapy may be enrolled and the use of antiplatelet is acceptable.

Exclusion Criteria:

* Any other severe acute or chronic medical or psychiatric condition besides the stroke.
* Women of child bearing potential.
* Uncontrolled hypertension.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (70):
- United States (32):
  - Spain Rehabilitation Center, Birmingham, Alabama
  - The Kirklin Clinic, Birmingham, Alabama
  - University Hospital, Birmingham, Alabama
  - Broward Health North, Deerfield Beach, Florida
  - Neurologic Consultant, P.A., Fort Lauderdale, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Neurostudies, Inc., Port Charlotte, Florida
  - Jagdish Sidhpura M.D., Columbus, Georgia
  - Jose Canedo, M.D., West Georgia Neurology, Columbus, Georgia
  - St. Francis Hospital, Columbus, Georgia
  - Muscogee Manor & Rehabilitation Center, Columbus, Georgia
  - Medical Research & Health Education Foundation, Inc., Columbus, Georgia
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Norwood Nursing Center, Huntington, Indiana
  - Massachusetts General Hospital/Department of Neurology, Boston, Massachusetts
  - Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Rehabilitation Institute of St. Louis, St Louis, Missouri
  - UNC HealthCare, Chapel Hill, North Carolina
  - UNC Department of Neurology Stroke Division, Chapel Hill, North Carolina
  - Investigational Drug Services at OU Medical Center, Oklahoma City, Oklahoma
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - OU Medical Center, Oklahoma City, Oklahoma
  - OU Physicians Building, Oklahoma City, Oklahoma
  - Penn State Milton South Hershey Medical Center / Penn State College of Medicine, Hershey, Pennsylvania
  - Penn State Hershey Rehabilitation Hospital, Hummelstown, Pennsylvania
  - The Methodist Hospital Neurological Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
- Bulgaria (7):
  - Voennomeditsinska Akademia - MBAL- Pleven, Otdelenie po Nervni bolesti, Pleven
  - MBAL Kaspela, Plovdiv
  - MBALNP "Sveti Naum" EAD, Klinika za Intenzivno Lechenie na Nervni Bolesti, Sofia
  - Vtora Mnogoprofilna Bolnitsa za Aktivno Lechenie, Otdelenie po Nevrologia, Sofia
  - MBAL "Tokuda Bolnitsa", Otdelenie po nevrologiya, Sofia
  - Universitetska mnogoprofilna bolnitsa za aktivno lechenie Aleksandrovska, Klinika po Nevrologia, Sofia
  - UMBAL Tsaritsa Yoanna, Klinika po nevrologia, Sofia
- Grey Nuns Community Hospital, Edmonton, Alberta, Canada
- Czechia (2):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Plzen, Plzen - Lochotin
- France (2):
  - CHU Pellegrin, Bordeaux
  - CHU La Pitie Salpetriere, Paris
- Germany (6):
  - Klinikum Altenburger Land, Altenburg
  - Universitaetsklinikum Essen, Neurologische Klinik, Essen
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum Rechts der Isar, Neurologische Klinik, München
  - Universitaetsklinikum Muenster, Münster
  - Universitaet Regensburg, Regensburg
- Hungary (6):
  - Dr. Kennessey Albert Korhaz-Rendelointezet, Neurologiai Osztaly, Balassagyarmat
  - Fovarosi Onkormanyzat Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont/Neurologia, Budapest
  - Semmelweis Egyetem AOK / Neurologiai Klinika, Budapest
  - Honvedkorhaz-Allami Egeszsegugyi Kozpont, Ideggyogyaszati Osztaly, Budapest
  - Orszagos Idegtudomanyi Intezet, Stroke-ambulancia, Budapest
  - Petz Aladar Megyei Oktato Korhaz, Neurologiai Osztaly, Győr
- India (2):
  - KEM Hospital, Pune, Maharashtra
  - Max Super Speciality Hospital, New Delhi
- South Korea (8):
  - Seoul National University Bundang Hospital, Department of Neurology, Seongnam-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Department of Neurology, Anyang-si, Gyonggi-do
  - Chonnam National University Hospital, Department of Neurology, Gwangju
  - Inha University Hospital, Department of Neurology, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Department of Neurology, Seoul
  - Samsung Medical Center, Department of Neurology, Seoul
  - Asan Medical Center, Department of Neurology, Seoul
- Taiwan (4):
  - Chang Gung Medical Foundation-Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan

REFERENCES:
- [Derived] Di Cesare F, Mancuso J, Woodward P, Bednar MM, Loudon PT; A9541004 Stroke Study Group. Phosphodiesterase-5 Inhibitor PF-03049423 Effect on Stroke Recovery: A Double-Blind, Placebo-Controlled Randomized Clinical Trial. J Stroke Cerebrovasc Dis. 2016 Mar;25(3):642-9. doi: 10.1016/j.jstrokecerebrovasdis.2015.11.026. Epub 2015 Dec 28. PMID 26738812
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9541004&StudyName=Study%20Evaluating%20The%20Safety%20And%20Efficacy%20Of%20PF-03049423%20In%20Subjects%20With%20Ischemic%20Stroke

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 181 participants were assigned to study treatment, 178 of which received study treatment.
Groups:
- Cohort 1: PF-03049423 1 mg: Participants received PF-03049423 1 mg once daily for 90 days.
- Cohort 1: Placebo: Participants received placebo matched to PF-03049423 1 mg once daily for 90 days.
- Cohort 2: PF-03049423 3 mg: Participants received PF-03049423 3 mg once daily for 90 days.
- Cohort 2: Placebo: Participants received placebo matched to PF-0304942 3 mg once daily for 90 days.
- Cohort 3: PF-03049423 6 mg: Participants received PF-03049423 6 mg once daily for 90 days.
- Cohort 3: Placebo: Participants received placebo matched to PF-0304942 6 mg once daily for 90 days.
Period: Overall Study
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Started | 11 | 9 | 11 | 10 | 70 | 67
Completed | 6 | 6 | 7 | 9 | 46 | 46
Not Completed | 5 | 3 | 4 | 1 | 24 | 21
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 3 | 5
Not completed — Death | 0 | 0 | 0 | 0 | 3 | 5
Not completed — Did not meet entrance criteria | 2 | 1 | 1 | 0 | 1 | 0
Not completed — Medication error without adverse event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 10 | 7
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Other | 2 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all randomized participants who took any study medication (active or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo | Total
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (14.3) | 64.7 (6.0) | 69.8 (8.3) | 65.8 (13.4) | 64.2 (13.1) | 65.6 (11.3) | 65.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 7 | 3 | 28 | 26 | 70
  Male | 7 | 7 | 4 | 7 | 42 | 41 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Abnormal Laboratory Test Results (Part 1* and 2)
Description: The total number of participants with laboratory test abnormalities (without regard to baseline abnormality) was assessed. *This endpoint was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for this timeframe were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 1 (Baseline) up to Day 90
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo). Participants analyzed indicated number of participants evaluated.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 10 | 10 | 70 | 66
participants | 8 | 8 | 10 | 9 | 64 | 56

2. Primary Outcome: Number of Participants With Vital Signs Data Met Criteria of Potential Clinical Concern (Part 1* and 2)
Description: Vital signs included blood pressure (BP; supine, sitting and standing) and pulse rate. Vital signs criteria of potential clinical concern were 1), BP: systolic BP (SBP) greater than or equal to (>=) 30 or 50 millimeters of mercury (mm Hg) change from grand baseline in same posture, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from grand baseline in same posture, diastolic <50 mm Hg; 2), pulse rate (supine, sitting and standing): <40 or greater than (>) 120 beats per minute (bpm); Standing: <40 or >140 bpm. *This endpoint was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for this timeframe were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 1 (Baseline) up to follow-up (28 days after Day 90)
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo). n=number of evaluable participants.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
participants
  Supine SBP <90 mm Hg, n=11,9,11,10,70,67 | 0 | 1 | 1 | 0 | 3 | 0
  Sitting SBP <90 mm Hg, n=10,8,9,5,55,59 | 0 | 1 | 1 | 0 | 2 | 2
  Standing SBP <90 mm Hg, n=7,7,9,8,49,48 | 0 | 0 | 0 | 0 | 1 | 1
  Supine DBP <50 mm Hg, n=11,9,11,10,70,67 | 0 | 0 | 2 | 1 | 6 | 4
  Sitting DBP <50 mm Hg, n=10,8,9,5,55,59 | 0 | 0 | 0 | 0 | 3 | 1
  Standing DBP <50 mm Hg, n=7,7,9,8,49,48 | 0 | 0 | 0 | 1 | 2 | 3
  Supine pulse rate <40 bpm, n=11,9,11,10,70,67 | 0 | 0 | 0 | 0 | 1 | 0
  Supine pulse rate >120 bpm, n=11,9,11,10,70,67 | 0 | 0 | 1 | 0 | 5 | 7
  Increase:supine SBP >=30 mm Hg, n=11,9,11,10,70,67 | 2 | 3 | 5 | 3 | 13 | 17
  Increase: sitting SBP >=30 mm Hg, n=9,6,9,4,48,44 | 0 | 2 | 2 | 0 | 10 | 9
  Increase: standing SBP >=30 mm Hg, n=2,3,3,6,19,22 | 0 | 0 | 0 | 2 | 2 | 1
  Increase:supine DBP >=20 mm Hg, n=11,9,11,10,70,67 | 4 | 2 | 5 | 2 | 16 | 22
  Increase: sitting DBP >=20 mm Hg, n=9,6,9,4,48,44 | 3 | 1 | 2 | 2 | 9 | 12
  Increase: standing DBP >=20 mm Hg, n=2,3,3,6,19,22 | 0 | 0 | 0 | 2 | 3 | 3
  Decrease:supine SBP >=30 mm Hg, n=11,9,11,10,70,67 | 7 | 6 | 5 | 4 | 37 | 37
  Decrease: sitting SBP >=30 mm Hg, n=9,6,9,4,48,44 | 3 | 4 | 6 | 2 | 26 | 18
  Decrease: standing SBP >=30 mm Hg, n=2,3,3,6,19,22 | 2 | 2 | 0 | 2 | 10 | 11
  Decrease:supine DBP >=20 mm Hg, n=11,9,11,10,70,67 | 8 | 6 | 6 | 3 | 32 | 26
  Decrease: sitting DBP >=20 mm Hg, n=9,6,9,4,48,44 | 1 | 4 | 5 | 1 | 23 | 14
  Decrease: standing DBP >=20 mm Hg, n=2,3,3,6,19,22 | 2 | 2 | 1 | 2 | 6 | 11
  Decrease:supine SBP >=50 mm Hg, n=11,9,11,10,70,67 | 2 | 0 | 1 | 2 | 10 | 9
  Decrease: sitting SBP >=50 mm Hg, n=9,6,9,4,48,44 | 2 | 1 | 3 | 0 | 7 | 6
  Decrease: standing SBP >=50 mm Hg, n=2,3,3,6,19,22 | 1 | 0 | 0 | 0 | 1 | 2
  Sitting pulse rate <40 bpm, n=1,0,2,0,3,2 | 0 | NA — No participants were evaluated. | 0 | NA — No participants were evaluated | 0 | 0
  Standing pulse rate <40 bpm, n=0,0,0,2,1,0 | NA — No participants were evaluated. | NA — No participants were evaluated. | NA — No participants were evaluated. | 0 | 0 | NA — No participants were evaluated.
  Sitting pulse rate >120 bpm, n=1,0,2,0,3,2 | 0 | NA — No participants were evaluated. | 0 | NA — No participants were evaluated. | 0 | 0
  Standing pulse rate >140 bpm, n=0,0,0,2,1,0 | NA — No participants were evaluated. | NA — No participants were evaluated. | NA — No participants were evaluated. | 0 | 0 | NA — No participants were evaluated.

3. Primary Outcome: Number of Participants With Electrocardiograms (ECGs) Data Met Criteria of Potential Clinical Concern (Part 1* and 2)
Description: ECG criteria of potential clinical concern were 1), PR interval: >=300 milliseconds (msec); >=25% increase when baseline >200 msec; or increase >=50% when baseline <=200 msec; 2), QRS interval: >=140 msec; >=50% increase from baseline; 3), QT interval: >=500 msec, QTc interval using Fridericia's formula (QTcF interval): absolute value >=450 - <480 msec, >=480-<500 msec, >=500 msec; absolute change 30 - <60, >=60 msec. *This endpoint was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for this timeframe were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 1 (Baseline) to Day 90
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
participants
  PR interval >=300 msec, n=11,9,11,10,70,67 | 0 | 0 | 0 | 0 | 0 | 0
  QRS interval >=140 msec, n=11,9,11,10,70,67 | 1 | 0 | 1 | 1 | 0 | 1
  QT interval >=500 msec, n=11,9,11,10,70,67 | 0 | 0 | 0 | 0 | 4 | 1
  QTcF interval 450-480 msec, n=11,9,11,10,70,67 | 2 | 3 | 4 | 2 | 14 | 14
  QTcF interval 480-500 msec, n=11,9,11,10,70,67 | 0 | 1 | 0 | 1 | 4 | 3
  QTcF interval >=500 msec, n=11,9,11,10,70,67 | 0 | 0 | 1 | 0 | 0 | 1
  PR interval increase >=25%/50%, n=10,7,9,9,52,47 | 0 | 0 | 1 | 0 | 1 | 0
  QRS interval increase >=50%, n=10,9,11,10,69,66 | 0 | 0 | 0 | 0 | 0 | 1
  QTcF increase 30-60 msec, n=10,9,11,10,69,66 | 2 | 3 | 4 | 2 | 19 | 11
  QTcF increase >=60 msec, n=10,9,11,10,69,66 | 0 | 0 | 0 | 1 | 3 | 5

4. Primary Outcome: Number of Participants With Significant Change in Physical Examination Findings (Part 1* and 2)
Description: The complete physical examination included examination of the skin, eyes, ears, throat, neck, cardiac, respiratory, gastrointestinal, and musculoskeletal systems. The limited physical examination included examination of the cardiac, respiratory, gastrointestinal, and musculoskeletal systems. *This endpoint was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for this timeframe were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 1 (Baseline) up to Day 90
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo). Participants analyzed indicated those who had physical examinations done at both baseline and last visit.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 66
participants | 1 | 1 | 0 | 0 | 2 | 0

5. Primary Outcome: Number of Participants With Significant Change in Neurological Examination Findings (Part 1* and 2)
Description: The complete neurological examination included an assessment of the motor, sensory, cranial nerves, reflexes, mental status and associated motor functions. The limited neurological exam could examine the same categories of neurologic assessments as the full examination, but would differ by the depth in the examination. The examination was required to be done to the extent needed to assess the participant for any potential changes in neurological status, as determined by the Investigator, but had to always include an assessment of motor, vision and hearing. *This endpoint was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for this timeframe were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 1 (Baseline) up to Day 90
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo). Participants analyzed indicated those who had neurological examinations done at both baseline and last visit.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 66
participants | 1 | 1 | 0 | 0 | 4 | 0

6. Primary Outcome: Number of Participants With Suicidal Behavior and/or Ideation as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) (Part 1* and 2)
Description: Data were mapped to Columbia-Classification Algorithm of Suicide Assessment (C-CASA) event codes. C-SSRS assessed if participant experienced: completed suicide (Code 1), suicide attempt (Code 2) (Response of "Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior (Code 3) ("Yes" on "aborted attempt", "interrupted attempt", "preparatory acts or behavior"), suicidal ideation (Code 4) ("Yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act/some intent to act without specific plan or with specific plan and intent), self-injurious behavior, no suicidal intent (Code 7) ("Yes" on "Has participant engaged in non-suicidal self-injurious behavior"). Number of participants with "Yes" response for any of above mentioned categories was assessed. *This was a primary endpoint for Part 1 (timeframe Days 1 to 14), as data for it were not reported separately, Part 1 and 2 data were reported together.
Time Frame: Day 7 (Baseline) up to follow up (28 days after Day 90)
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo). n=number of participants who had C-SSRS assessed at that visit.
Measure: Number; unit: participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
participants
  Day 7, n=0, 0, 1, 1, 64, 57 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 1 | 2
  Day 14, n=0, 0, 1, 1, 59, 53 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 1 | 0
  Day 30, n=0, 0, 1, 1, 60, 47 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 2 | 0
  Day 60, n=0, 0, 1, 1, 55, 44 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 2 | 0
  Day 90, n=0, 0, 1, 1, 61, 53 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 1 | 1
  Follow-up, n=0, 0, 1, 1, 59, 51 | NA — No participants had C-SSRS assessed. | NA — No participants had C-SSRS assessed. | 0 | 0 | 0 | 0

7. Primary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Less Than or Equal to (<=2) at Day 90 (Part 2)
Description: The mRS is a 6-point scale of functional recovery. The scale grades participants as having no symptoms (0), minor symptoms (1), minor handicap (2), moderate handicap (3), moderately severe handicap (4), severe handicap (5), or death (6).
Time Frame: Day 90
Population: The Inferential Full Analysis Set (I-FAS) consisted of participants within the FAS who were randomized to PF-03049423 maximum tolerated dose (MTD) or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). n=number of participants included for comparison between active drug and placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants
  Last Observation Carried Forward (LOCF), n=68, 65 | 42.6 | 46.2
  Observed Cases (OC), n=51, 52 | 47.1 | 50.0
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.4962, Regression, Logistic; LOCF was used to impute missing data; Odds Ratio (OR) = 0.735, 80% CI 2-sided [0.41 to 1.31]
Statistical Analysis 2: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.2517, Regression, Logistic; The analysis was based on OC; Odds Ratio (OR) = 0.561, 80% CI 2-sided [0.29 to 1.07]

8. Secondary Outcome: Change From Baseline in Box and Blocks (B&B) Test at Day 90 for Paretic Hand (Part 2)
Description: The B&B test is a measure of manual dexterity. The B&B apparatus consists of a box divided into 2 sections and 1-inch hardwood blocks. The blocks began in the compartment of the test box to the dominant side of the participant. The participant was required to transfer the blocks one at a time to the other side of the box as quickly as possible in 1 minute using the non-paretic hand. The box was then turned so all the blocks were in the same side as the paretic hand. The participant was then required to do the test with his/her paretic hand. The participant was told that if more than 1 block was picked up at a time it was to only count as 1 block. The participant was also told that their fingertips needed to cross the partition for the block to be counted. The performance measure for this task was the number of blocks moved within 1 minute.
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). Number of participants indicated those participants included for comparison between active drug and placebo.
Measure: Least Squares Mean (Standard Error); unit: blocks moved per minute
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 21 | 24
blocks moved per minute | 26.881 (3.8667) | 26.741 (3.5627)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Paretic hand; Test type: Superiority or Other; p = 0.9716, Mixed Models Analysis; Mean Difference (Final Values) = 0.141, 80% CI 2-sided [-4.972 to 5.254], Standard Error of Mean 3.9420

9. Secondary Outcome: Change From Baseline in Box and Blocks (B&B) Test at Day 90 for Paretic to Non-paretic Hand Ratio (Part 2)
Description: as for outcome 8
Time Frame: Day 1 (Baseline), Day 90
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 21 | 24
percentage change | 41.830 (7.7810) | 31.041 (7.1284)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Paretic to non-paretic hand ratio (%); Test type: Superiority or Other; p = 0.1417, Mixed Models Analysis; Mean Difference (Final Values) = 10.789, 80% CI 2-sided [1.401 to 20.177], Standard Error of Mean 7.2392

10. Secondary Outcome: Change From Baseline in Hand Grip Strength Test at Day 90 for Paretic and Non-paretic Hands (Part 2)
Description: The Hand Grip Strength Test measures the maximum isometric strength of the hand and forearm muscles. The participant was required to squeeze the dynamometer with maximum isometric effort while sitting with shoulder adducted and neutrally roated, elbow flexed at 90 degrees and the forearm in neutral position and wrist between 0 to 30 degrees dorsiflexion and a 0 to 15 degrees ulnar deviation. The participant performed this task 3 times with each hand, starting with the non-paretic hand. The performance measure for this task was the average score measured in pounds of pressure exerted.
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). n=number of participants included for comparison between active drug and placebo.
Measure: Least Squares Mean (Standard Error); unit: pounds
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
pounds
  Paretic Hand, n=26, 26 | 20.556 (4.1829) | 30.886 (3.9964)
  Non-Paretic Hand, n=46, 41 | 12.546 (2.3612) | 12.312 (2.5029)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Paretic hand; Test type: Superiority or Other; p = 0.0611, Mixed Models Analysis; Mean Difference (Final Values) = -10.330, 80% CI 2-sided [-17.351 to -3.310], Standard Error of Mean 5.4241
Statistical Analysis 2: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Non-paretic hand; Test type: Superiority or Other; p = 0.9433, Mixed Models Analysis; Mean Difference (Final Values) = 0.235, 80% CI 2-sided [-4.011 to 4.480], Standard Error of Mean 3.2899

11. Secondary Outcome: Change From Baseline in Hand Grip Strength Test at Day 90 for Paretic to Non-paretic Hand Ratio (Part 2)
Description: as for outcome 10
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). Number of participants analyzed indicated those participants included for comparison between active drug and placebo.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 26 | 26
percentage change | 23.949 (5.4499) | 36.761 (5.1182)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Paretic to non-paretic hand ratio (%); Test type: Superiority or Other; p = 0.0654, Mixed Models Analysis; Mean Difference (Final Values) = -12.812, 80% CI 2-sided [-21.668 to -3.957], Standard Error of Mean 6.8448

12. Secondary Outcome: Percentage of Participants With mRS (0-1) at Day 90 (Part 2)
Description: as for outcome 7
Time Frame: Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants | 25.0 | 24.6
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; LOCF was used to impute missing data; Test type: Superiority or Other; p = 0.9510, Regression, Logistic; Odds Ratio (OR) = 0.972, 80% CI 2-sided [0.54 to 1.76]

13. Secondary Outcome: Percentage of Participants With National Institutes of Health Stroke Scale (NIHSS) (0-1) at Day 90 (Part 2)
Description: The NIHSS is a graded 11-item neurological examination rating speech and language, cognition, visual field deficits, motor and sensory impairments and ataxia used for the clinical assessment of acute stroke therapy. The maximum total score is 42 in a participant with a severe neurological deficit; the minimum score is 0 in a participant without gross neurological deficits.
Time Frame: Day 90
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants | 25.0 | 26.2
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; LOCF was used to impute missing data; Test type: Superiority or Other; p = 0.7234, Regression, Logistic; Odds Ratio (OR) = 0.854, 80% CI 2-sided [0.48 to 1.51]

14. Secondary Outcome: Change From Baseline in NIHSS at Day 90 (Part 2)
Description: as for outcome 13
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). Participants analyzed indicated number of participants included for comparison between active drug and placebo for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 47
unit on a scale | -6.511 (0.5384) | -6.228 (0.5655)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.6759, Mixed Models Analysis; Mean Difference (Final Values) = -0.283, 80% CI 2-sided [-1.156 to 0.589], Standard Error of Mean 0.6755

15. Secondary Outcome: Percentage of Participants With Barthel Index (BI) >= 95 and BI =100 at Day 90 (Part 2)
Description: The BI is an index of independence to score the ability of a participant with a neuromuscular or musculoskeletal disorder to care for him or herself. The index rates a participant's ability on the following 10 activities: feeding, moving from wheelchair to bed, personal toilet, getting on and off toilet, bathing self, walking on level surface, ascending and descending stairs, dressing, controlling bowels and controlling bladder. The maximum total score is 100 in a participant without functional impairment; the minimum score is 0 in a participant with major functional impairment.
Time Frame: Day 90
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants
  BI >=95 | 47.1 | 40.0
  BI=100 | 42.6 | 35.4
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; BI >=95, LOCF was used to impute missing data; Test type: Superiority or Other; p = 0.4213, Regression, Logistic; Odds Ratio (OR) = 1.433, 80% CI 2-sided [0.81 to 2.54]
Statistical Analysis 2: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; BI=100, LOCF was used to impute missing data; Test type: Superiority or Other; p = 0.2760, Regression, Logistic; Odds Ratio (OR) = 1.651, 80% CI 2-sided [0.92 to 2.98]

16. Secondary Outcome: BI at Day 90 (Part 2)
Description: as for outcome 15
Time Frame: Day 90
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: unit on a scale
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 49 | 47
unit on a scale | 79.151 (3.6248) | 73.552 (3.8471)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.2118, Mixed Models Analysis; Mean Difference (Final Values) = 5.599, 80% CI 2-sided [-0.150 to 11.348], Standard Error of Mean 4.4547

17. Secondary Outcome: Domains of Interest: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Coding Sub Test at Day 90 (Part 2)
Description: The test uses a reference key, the participant had 90 seconds to pair specific numbers with given geometric figures. Responses could be written or oral. The performance measure for this task was the total number of correct responses.
Time Frame: Day 1 (Baseline), Day 90
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: correct responses
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 33 | 28
correct responses | 13.748 (1.5321) | 12.686 (1.6282)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.5541, Mixed Models Analysis; Mean Difference (Final Values) = 1.062, 80% CI 2-sided [-1.252 to 3.375], Standard Error of Mean 1.7844

18. Secondary Outcome: Domains of Interest: Change From Baseline in RBANS Naming Sub Test at Day 90 (Part 2)
Description: This test requires the participant to name 10 objects drawn in ink. The tester asked the participant to identify the picture. The participant had 20 seconds to respond to each picture presented. The performance measure was the number of objects named correctly.
Time Frame: Day 1 (Baseline), Day 90
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: objects named correctly
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 41 | 37
objects named correctly | 0.989 (0.3676) | 1.324 (0.3666)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.4260, Mixed Models Analysis; Mean Difference (Final Values) = -0.334, 80% CI 2-sided [-0.874 to 0.205], Standard Error of Mean 0.4178

19. Secondary Outcome: Domains of Interest: Change From Baseline in Line Cancellation Test [(L+R)/28 × 100%, (L/14) × 100%, (R/14) × 100%)] at Day 90 (Part 2)
Description: The participant was presented with a page that had lines placed across the page. The participant was required to cross out all the lines on the page using their non-paretic hand after the tester had demonstrated what was required by crossing out the center line. The performance measure for this task was the total number of omissions made expressed as a percentage of the total number of items in the test. The test contains 4 variables: (L+R)/28 × 100%, (L/14) × 100%, (R/14) × 100%, and (L-R)/(L+R), where L = number of lines crossed on the left side of the paper; R = number of lines crossed on the right side of the paper.
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). n=number of participants included for comparison between active drug and placebo for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: change in percentage of lines crossed
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 68 | 65
change in percentage of lines crossed
  (L+R)/28 × 100%, n=39, 35 | 19.459 (4.4433) | 16.983 (4.4551)
  (L/14) × 100%, n=39, 35 | 22.824 (5.6691) | 18.950 (5.6639)
  (R/14) × 100%, n=39, 35 | 16.481 (4.3564) | 15.431 (4.3647)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; (L+R)/28 × 100%; Test type: Superiority or Other; p = 0.6500, Mixed Models Analysis; Mean Difference (Final Values) = 2.477, 80% CI 2-sided [-4.547 to 9.500], Standard Error of Mean 5.4394
Statistical Analysis 2: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; (L/14) × 100%; Test type: Superiority or Other; p = 0.5671, Mixed Models Analysis; Mean Difference (Final Values) = 3.874, 80% CI 2-sided [-4.834 to 12.583], Standard Error of Mean 6.7431
Statistical Analysis 3: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; (R/14) × 100%; Test type: Superiority or Other; p = 0.8430, Mixed Models Analysis; Mean Difference (Final Values) = 1.049, 80% CI 2-sided [-5.771 to 7.870], Standard Error of Mean 5.2816

20. Secondary Outcome: Domains of Interest: Change From Baseline in Line Cancellation Test at Day 90 [(L-R)/(L+R)] (Part 2)
Description: as for outcome 19
Time Frame: Day 1 (Baseline), Day 90
Population: The I-FAS consisted of participants within the FAS who were randomized to PF-03049423 MTD or highest dose (6 mg) group or the placebo group that was in the same cohort as the MTD or highest dose (6 mg). Number of participants analyzed indicated participants included for comparison between active drug and placebo for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: change in ratio
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 39 | 34
change in ratio | 0.083 (0.0620) | -0.023 (0.0625)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; (L R)/(L+R); Test type: Superiority or Other; p = 0.1512, Mixed Models Analysis; Mean Difference (Final Values) = 0.106, 80% CI 2-sided [0.011 to 0.201], Standard Error of Mean 0.0733

21. Secondary Outcome: Domains of Interest: Change From Baseline in Recognition Memory Test at Day 90 (Part 2)
Description: This test assesses the ability to recognize pictures of objects. The participant was presented a series of pictures, a subset of which were the objects presented in the RBANS Naming Sub Test. After each picture was presented, the participant indicated either manually (ie, affirmative head nod) or verbally whether the picture was seen previously. The participant was given 5 seconds per picture to respond. The performance measure for this task was the total number of pictures correctly identified.
Time Frame: Day 1 (Baseline), Day 90
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: pictures correctly identified
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 44 | 37
pictures correctly identified | -1.135 (0.4743) | 0.144 (0.4797)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.0128, Mixed Models Analysis; Mean Difference (Final Values) = -1.279, 80% CI 2-sided [-1.929 to -0.629], Standard Error of Mean 0.5041

22. Secondary Outcome: Gait Velocity Test at Day 90 (Part 2)
Description: The 10-meter walk test requires a 20 meter straight path, with 5 meters for acceleration, 10 meters for steady state walking, and 5 meters for deceleration. Markers were placed at the 5 and 15 meter positions along the path. The participant began to walk "at a comfortable pace" at 1 end of the path, and continued walking until he/she reached the other end. The rater used a stopwatch to determine how much time it took for the participant to traverse the 10 meter center of the path, starting the stopwatch as soon as the participant's limb crossed the first marker and stopping the stopwatch as soon as the participant's limb crossed the second marker.
Time Frame: Day 90
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: meters/second (m/s)
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 41 | 36
meters/second (m/s) | 1.064 (0.1040) | 0.975 (0.1128)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Test type: Superiority or Other; p = 0.4713, Mixed Models Analysis; Mean Difference (Final Values) = 0.089, 80% CI 2-sided [-0.070 to 0.248], Standard Error of Mean 0.1226

23. Secondary Outcome: Plasma Concentrations of PF-03049423 (Part 1 and 2)
Time Frame: Days 1, 2, 7, 14, 30, 60 and 90
Population: PK concentration population included all participants who were treated with PF-03049423 who had at least 1 measurable concentration. n=participants with concentration above lower limit of quantification at the corresponding sampling time.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 2: PF-03049423 3 mg | Cohort 3: PF-03049423 6 mg
Number analyzed (Participants) | 11 | 11 | 70
nanogram/milliliter (ng/mL)
  Day 1 (0 hour predose), n=0, 1, 3 | NA (NA) — No participants had concentration above lower limit quantification. | 0.05245 (0.17397) | 1.420 (11.591)
  Day 1 (1 hour post dose), n=11, 10, 63 | 5.825 (4.3514) | 17.50 (12.814) | 46.76 (36.153)
  Day 1 (2 hours post dose), n=11, 11, 61 | 7.063 (3.2729) | 30.18 (11.313) | 58.19 (32.837)
  Day 1 (8 hours post dose), n=11, 11, 68 | 7.361 (2.4032) | 25.39 (8.6644) | 52.47 (23.250)
  Day 2 (0 hour, predose), n=11, 11, 67 | 4.521 (1.5265) | 18.05 (4.7834) | 32.07 (13.776)
  Day 7 (0 hour, post dose), n=9, 7, 64 | 8.601 (2.9609) | 27.79 (7.6945) | 53.08 (30.237)
  Day 7 (1 hour post dose), n=0, 1, 59 | NA (NA) — No samples were collected. | 51.80 (NA) — 1 participant had concentration above lower limit of quantification, SD cannot be calculated. | 115.9 (65.329)
  Day 7 (2 hours post dose), n=0, 1, 59 | NA (NA) — No samples were collected. | 58.10 (NA) — 1 participant had concentration above lower limit of quantification, SD cannot be calculated. | 126.3 (57.759)
  Day 7 (6 hours post dose), n=0, 1, 61 | NA (NA) — No samples were collected. | 51.10 (NA) — 1 participant had concentration above lower limit of quantification, SD cannot be calculated. | 103.8 (41.090)
  Day 14 (0 hour predose), n=10, 8, 59 | 7.805 (2.9278) | 31.13 (9.8243) | 53.10 (28.085)
  Day 14 (1 hour post dose), n=9, 7, 0 | 16.47 (7.1782) | 76.71 (32.657) | NA (NA) — No samples were collected.
  Day 14 (2 hours post dose), n=9, 6, 0 | 17.06 (7.3799) | 70.37 (14.795) | NA (NA) — No samples were collected.
  Day 14 (6 [cohort 3:4] hours post dose), n=9,7,31 | 17.57 (4.1614) | 58.36 (11.720) | 118.2 (41.967)
  Day 30 (0 hour predose), n=6, 6, 58 | 5.339 (3.5712) | 29.68 (11.015) | 50.77 (31.473)
  Day 30 (4 hours post dose), n=2, 5, 25 | 11.55 (2.6234) | 57.08 (13.990) | 96.27 (49.929)
  Day 60 (0 hour predose), n=6, 6, 53 | 6.360 (3.1028) | 24.55 (5.8206) | 49.37 (33.747)
  Day 60 (4 hours post dose), n=2, 5, 27 | 13.25 (0.7778) | 47.86 (7.3296) | 112.1 (58.560)
  Day 90 (0 hour predose), n=5, 6, 45 | 5.252 (1.5161) | 29.18 (15.909) | 47.02 (24.065)
  Day 90 (4 hours post dose), n=2, 5, 20 | 12.80 (0.000) | 49.40 (13.962) | 82.69 (29.005)

24. Other Pre Specified Outcome: All-cause Mortality (Part 2)
Description: Deaths regardless causality were reported.
Time Frame: The time began from the participant provided informed consent through 28 calendar days post last administration of investigational product.
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo).
Measure: Number; unit: Number of participants
Groups:
- Cohort 2: Placebo: Participants received placebo matched to PF-03049423 3 mg once daily for 90 days.
- Cohort 3: Placebo: Participants received placebo matched to PF-03049423 6 mg once daily for 90 days.
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
Number of participants | 0 | 0 | 0 | 0 | 6 | 7

25. Other Pre Specified Outcome: Mortality Directly Related to Stroke (Part 2)
Description: Deaths caused by stroke were reported.
Time Frame: as for outcome 24
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo).
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
Number of participants | 0 | 0 | 0 | 0 | 3 | 0

26. Other Pre Specified Outcome: Number of Participants With Neuro-worsening (Part 2)
Description: NIHSS change of 4 points or greater.
Time Frame: Day 1 (Baseline) up to Day 90
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo).
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
Number of participants | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of NIHSS data.

27. Other Pre Specified Outcome: Number of Participants With SBP <100 mm Hg or SBP Decline >=30 mm Hg From Immediate Pre-dose Measurement, With or Without Neuro-worsening (Defined as an NIHSS Increase of 4 Points or Greater) Within 2 Hours Post-dose (Part 2)
Time Frame: Day 1 (Baseline) up to Day 14
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo).
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
Number of participants | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data. | NA — No data were reported separately for this outcome measure, which was instead included in routine clinical review of BP data.

28. Other Pre Specified Outcome: Treatment-emergent Adverse Events (AEs) Resulting in Discontinuation of Study Drug (Part 2)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 (Baseline) up to follow-up (28 days after Day 90)
Population: The FAS consisted of all randomized participants who took any study medication (active or placebo).
Measure: Number; unit: Number of participants
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 11 | 9 | 11 | 10 | 70 | 67
Number of participants | 0 | 1 | 2 | 0 | 3 | 5

29. Secondary Outcome: Change From Baseline in Box and Blocks (B&B) Test at Day 90 for Non-paretic Hand (Part 2)
Description: as for outcome 8
Time Frame: Day 1 (Baseline), Day 90
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: blocks moved per minute
Arm/Group | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Number analyzed (Participants) | 45 | 41
blocks moved per minute | 17.797 (2.1676) | 18.313 (2.2407)
Statistical Analysis 1: Comparison: Cohort 3: PF-03049423 6 mg vs Cohort 3: Placebo; Non-paretic hand; Test type: Superiority or Other; p = 0.8501, Mixed Models Analysis; Mean Difference (Final Values) = -0.516, 80% CI 2-sided [-4.026 to 2.995], Standard Error of Mean 2.7201

ADVERSE EVENTS:
Time Frame: From the time the subject had taken at least 1 dose of study treatment through last subject visit. For SAEs, the time began from the subject provided informed consent through 28 calendar days post last administration of investigational product.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Cohort 1: PF-03049423 1 mg | Cohort 1: Placebo | Cohort 2: PF-03049423 3 mg | Cohort 2: Placebo | Cohort 3: PF-03049423 6 mg | Cohort 3: Placebo
Serious Adverse Events (participants affected / at risk) | 2/11 | 1/9 | 3/11 | 1/10 | 15/70 | 18/67
Other Adverse Events (participants affected / at risk) | 10/11 | 7/9 | 7/11 | 9/10 | 50/70 | 47/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-03049423 1 mg (N=11) | Cohort 1: Placebo (N=9) | Cohort 2: PF-03049423 3 mg (N=11) | Cohort 2: Placebo (N=10) | Cohort 3: PF-03049423 6 mg (N=70) | Cohort 3: Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-03049423 1 mg (N=11) | Cohort 1: Placebo (N=9) | Cohort 2: PF-03049423 3 mg (N=11) | Cohort 2: Placebo (N=10) | Cohort 3: PF-03049423 6 mg (N=70) | Cohort 3: Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 4 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 2 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 2 | 0 | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 2 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 8 | 14
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 2 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 4
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 3 | 3
Pyrexia (General disorders) | 1 | 0 | 2 | 0 | 7 | 6
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 8 | 8
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 2 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 3
Aspartate aminotransferase abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 4
Blood bilirubin abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 7 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 9 | 4
Dementia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 3
Haemorrhagic transformation stroke (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 3 | 1 | 0 | 5 | 7
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 2
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 5 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 4 | 4
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 7 | 2
Sleep disorder (Psychiatric disorders) | 3 | 0 | 0 | 0 | 4 | 1
Albuminuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 5 | 4
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 7 | 2
Renal cyst (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 2
Urethral haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 4 | 0 | 1 | 3 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 4 | 7

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to demonstrated futility at interim analysis. The final results are consistent with interim results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.